CLINICAL TRIAL: NCT07377643
Title: A Randomized, Multicenter, Open-label Phase 3 Study to Compare IBI354 With or Without Pertuzumab vs. Taxane in Combination With Trastuzumab and Pertuzumab as First-line Treatment in Participants With Unresectable, Locally Advanced or Metastatic HER2-Positive Breast Cancer
Brief Title: IBI354 With or Without Pertuzumab Versus Taxane, Trastuzumab and Pertuzumab in HER2-positive Metastatic Breast Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Innovent Biopharmaceutical Technology (Hangzhou) Co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIBI354B302
Record Dates: First submitted 2026-01-15; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: HER2-positive Breast Cancer
MeSH Terms: interventions — Trastuzumab; Docetaxel; pertuzumab; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): IBI354 plus pertuzumab
  Interventions: Drug: IBI354; Drug: Pertuzumab
- Group C (Active Comparator): THP
  Interventions: Drug: Trastuzumab; Drug: Docetaxel; Drug: Pertuzumab; Drug: Paclitaxel
- Group B (Experimental): IBI354
  Interventions: Drug: IBI354

INTERVENTIONS:
Drug: Trastuzumab — IV infusion
  Arms: Group C
Drug: IBI354 — IV infusion
  Arms: Group A; Group B
Drug: Docetaxel — IV infusion
  Arms: Group C
Drug: Pertuzumab — IV infusion
  Arms: Group A; Group C
Drug: Paclitaxel — IV infusion
  Arms: Group C

SUMMARY:
This is a randomized, multicenter, open-label, phase 3 study evaluating the efficacy, safety, and tolerability of IBI354 combined with or without pertuzumab vs. THP as first-line treatment for HER2-positive unresectable, locally advanced or metastatic breast cancer.

ELIGIBILITY:
Participants are eligible to be included in the study only if they meet all of the following criteria:

1. Have signed the informed consent form (ICF) and are able to comply with the follow-up visits and related procedures required in the protocol.
2. Male or female participants: ≥18 years of age
3. Pathologically confirmed breast cancer:

   1. Unresectable, locally advanced or metastatic breast cancer, i.e. participants who cannot be treated with curative intent and confirmed HER2-positive (HER2 IHC 3+ or HER2 ISH+) on specimens taken after confirmed locally advanced or metastatic disease by central testing.
   2. Documented history of hormone receptor (HR)-positive (defined as estrogen receptor [ER] and/or progesterone receptor [PgR] positive [ER or PgR ≥1%]) or HR-negative after local testing in the metastatic setting according to ASCO/CAP guidelines. If a participant has more than one ER/PgR result after metastatic disease, the most recent result will be used.
4. No prior chemotherapy or HER2-targeted therapy for unresectable, locally advanced or metastatic breast cancer (first-line endocrine therapy is allowed for patients with metastatic breast cancer). Participants who have received chemotherapy or HER2-directed therapy in the neoadjuvant or adjuvant therapies and have a DFI of >6 months from completion of systemic chemotherapy or HER2-targeted therapy to advanced or metastatic diagnosis are eligible.
5. Eastern Cooperative Oncology Group Performance Status (ECOG PS) score of 0 or 1.
6. Evidence of radiographic or objective disease progression on or after the last systemic therapy prior to starting study treatment.
7. Have a life expectancy of ≥12 weeks at screening.
8. At least 1 measurable lesion as defined per RECIST v1.1 that has not been previously irradiated. Must be ≥ 10 mm in long axis (except for lymph nodes, which must be ≥ 15 mm in short axis) when accurately measured at baseline by CT or MRI (preferably with intravenous contrast) and the lesion is suitable for repeated accurate measurement.
9. Left ventricular ejection fraction (LVEF) ≥ 50% within 28 days prior to randomization.
10. Adequate organ and bone marrow function. Laboratory test values within 7 days prior to the first dose of the investigational product meet the following requirements in (if the laboratory tests during the screening period do not meet the following requirements, only one retest is allowed during the screening period):

    1. Hemoglobin (HGB) ≥ 90 g/L (transfusion of red blood cells or erythropoietin are not allowed within 1 week prior to the screening assessment, and participants requiring ongoing transfusion or growth factor support to maintain hemoglobin ≥ 90 g/L are not eligible).
    2. Absolute neutrophil count (ANC) ≥ 1.5 × 109 /L or within the normal range (G-CSF is not allowed within 1 week prior to the screening assessment).
    3. Platelet (PLT) ≥ 90 × 109 /L (transfusion with platelets or thrombopoietin is not allowed within 1 week prior to screening assessment, participants requiring thrombopoietic growth factors to maintain adequate platelet count are not eligible).
    4. Total bilirubin (TBIL) ≤ 1.5 × upper limit of normal (ULN) in the absence of liver metastasis; TBIL < 3 × ULN in the presence of Gilbert syndrome (unconjugated hyperbilirubinemia) or liver metastasis.
    5. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3×ULN (<5×ULN for participants with liver metastases).
    6. Serum albumin ≥ 25 g/L.
    7. Serum creatinine ≤ 1.5 × ULN, or creatinine clearance ≥ 60 mL/min ( calculated using the Cockcroft-Gault formula ); if urinalysis indicates that the urine protein is < 2+, participants with urine protein ≥ 2+ from urinalysis at baseline should undergo a 24-hour urine collection and have a 24-hour urine protein quantitation < 1 g (if both methods are used, a 24-hour urine protein quantitation will be used to determine participant eligibility). Cockcroft/Gault formula:

       Female: CrCl = (140 - Age) × Weight (kg) × 0.85 72 × serum creatinine (mg/dL) Male: CrCl = (140 - years) × weight (kg) × 1.00 72 × serum creatinine (mg/dL)
    8. International normalized ratio (INR) ≤ 1.5 × ULN, and prothrombin time (PT) or activated partial thromboplastin time (APTT) ≤ 1.5 × ULN.
11. Participants with evidence of postmenopausal status or negative serum pregnancy test (Sexually active, WOCBP with a non-sterilized male partner) must have a negative serum pregnancy test at the screening visit. WOCBP are women who are not surgically sterile (i.e., have undergone bilateral salpingectomy, bilateral oophorectomy, or total hysterectomy) or are not postmenopausal.
12. Female participants of childbearing potential or male participants with partners of childbearing potential must take effective contraceptive measures during the entire course of the trial and 6 months after the treatment

Participants should not be included in the study if they meet any of the following criteria:

1. Prior treatment with antibody-drug conjugates containing camptothecin or its derivatives (topoisomerase I inhibitors).
2. Uncontrolled or significant cardiovascular and cerebrovascular diseases, including any of the following:

   1. History of myocardial infarction or symptomatic congestive heart failure (New York Heart Association [NYHA] class II to IV) or uncontrolled myocarditis within 6 months before randomization. Participants with troponin levels above the ULN at screening (as specified by the manufacturer) and without any myocardial infarction-related symptoms should have a cardiology consultation before randomization to rule out myocardial infarction.
   2. Uncontrolled hypertension (systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg) despite of standard treatment.
   3. History of any arterial thromboembolic events within 6 months prior to randomization, including myocardial infarction, unstable angina, cerebrovascular accident, or transient ischemic attack.
   4. History of deep vein thrombosis, pulmonary embolism, or any other serious thromboembolic events within 3 months prior to randomization (thrombosis or catheter-derived thrombosis of caused by implanted venous ports, or superficial vein thrombosis, intermuscular vein thrombosis are not considered serious thromboembolisms).
   5. History of arrhythmia (polymorphic premature ventricular contractions, bigeminy, trigeminy, ventricular tachycardia, ventricular fibrillation, torsades de pointes) that is symptomatic or requires treatment (CTCAE 5.0 Grade 3), atrial fibrillation that is symptomatic or uncontrolled despite treatment, or asymptomatic sustained ventricular tachycardia. Participants whose atrial fibrillation is controlled by medication or whose arrhythmia is controlled by a pacemaker will be allowed to be enrolled in the study.
   6. Fridericia-corrected QT interval (QTcF) >480 msec. If QTcF is > 480 ms in 1 ECG during the screening period, 3 consecutive ECGs should be performed and the mean QTcF should be calculated. If QTcF is still > 480 ms, the participant will not be enrolled.
   7. History of QT prolongation associated with other drugs that require discontinuation, or any current concomitant medication known to prolong QT interval leading to Torsade de Pointes.
   8. Congenital long QT syndrome, family history of long QT syndrome, or unexplained sudden death in first-degree relatives under 40 years old.
3. Non-infectious pneumonitis that requires corticosteroid treatment, or other clinically significant lung diseases such as a history of interstitial lung disease (ILD)/non-infectious pneumonitis, current ILD/non-infectious pneumonitis, or uncontrolled lung diseases (e.g., pulmonary fibrosis, severe radiation pneumonitis, and acute lung injury) or suspected ILD/non-infectious pneumonitis cannot be ruled out by imaging at screening.
4. Have a lung-specific intercurrent clinically significant illness including, but not limited to, any underlying pulmonary disorder (e.g., pulmonary embolism within 3 months prior to study randomization, severe asthma, severe chronic obstructive pulmonary disease [COPD], restrictive lung disorder, significant pleural effusion, post-COVID-19 pulmonary fibrosis, etc.), and any autoimmune, connective tissue, or inflammatory disorder with pulmonary involvement (or suspected at screening for pulmonary involvement) (e.g., rheumatoid arthritis, Sjogren's syndrome/Sjogren's syndrome, sarcoidosis etc.), and/or prior pneumonectomy.
5. Prior to the first dose of study drug:

   1. Antibody-based anticancer therapy within 4 weeks, except for receptor activator of nuclear factor-κb ligand (RANKL) inhibitors (eg, denosumab for the treatment of complications resulting from bone metastases).
   2. Hormonal therapy or immunotherapy (based on non-antibody therapy) within 3 weeks.
   3. Fixed-field palliative radiotherapy within 2 weeks, or wide-field palliative radiotherapy within 4 weeks or palliative radiotherapy cumulatively exceeding 30% of bone marrow.
   4. Received oral chemotherapy drugs, small molecule targeted drugs, and Chinese herbal medicines indicated for anti-tumor treatment within 2 weeks or 5 half-lives (whichever is longer).
   5. Had major surgery (craniotomy, thoracotomy, or laparotomy, and other types of surgery considered "major" by the investigator, excluding needle biopsy and vascular access) or major traumatic injury within 4 weeks, or expected major surgery during the study, or with severe unhealed wounds, trauma, or ulcers.
   6. Treatment with strong inhibitors or inducers of cytochrome P450 3A4 (CYP3A4) within 2 weeks or 5 half-lives (whichever is longer).
   7. Live vaccines (mRNA and non-replicating adenovirus vaccines are not considered live) within 4 weeks.
6. Participants who had used immunosuppressive medications within 14 days prior to the first dose of study drug, with the exception of intranasal and inhaled corticosteroids or systemic corticosteroids at doses of less than 10 mg/day prednisone (or equivalent to 10 mg/day prednisone) or for prevention of contrast dye allergy.
7. Known symptomatic central nervous system (CNS) metastasis and/or spinal cord compression and/or carcinomatous meningitis, or a history of leptomeningeal carcinoma. Participants with asymptomatic CNS metastases (without neurological symptoms, without the need for corticosteroids or anticonvulsants, and with metastases all ≤ 1.5 cm in diameter) or with brain metastases that are stable after treatment and meet all of the following criteria may be considered for inclusion: (1) measurable lesions outside the CNS; (2) no midbrain, pons, cerebellum, meninges, medulla oblongata, or spinal cord metastases; (3) stable for at least 4 weeks with no new or enlarging metastases ( clearly confirmed by clinical symptoms, signs, and imaging evidence); (4) have discontinued corticosteroids and/or anticonvulsants for at least 2 weeks prior to the first dose of study drug and have recovered from the acute toxicity of radiotherapy. Whole brain radiotherapy or stereotactic radiotherapy must be completed at least 2 weeks prior to study randomization. CNS lesions should be monitored and examined regularly during the study.

   Note: CNS lesions will not be considered target lesions.
8. Non-remission of adverse events (AEs) after previous anti-cancer treatment, defined as AEs that have not been relieved to ≤ grade 1 or baseline before enrollment according to NCI-CTCAE v5.0 criteria (except for alopecia and pigmentation). Note: Participants with chronic, stable Grade 2 toxicities (defined as not worsening to >Grade 2 for at least 3 months prior to enrollment and manageable with standard of care) that were considered by the investigator to be related to prior anticancer therapy, e.g., fatigue, insomnia, hypomagnesemia, chemotherapy-induced peripheral neuropathy, hypothyroidism stably controlled by replacement therapy, and hypertension stably controlled below 160/100 mmHg by antihypertensives, were eligible for study entry.
9. Tumor invades surrounding important tissues and organs (such as mediastinal great vessels, superior vena cava and inferior vena cava, pericardium, heart, trachea, esophagus, etc.).
10. Bleeding within 3 months prior to the first dose of study treatment that is life-threatening and requires blood transfusion or invasive treatment.
11. Symptomatic abdominopelvic fluid collections, pleural effusions, or pericardial effusions requiring intervention (participants with stable controlled effusions, defined as clinically asymptomatic effusions that do not increase significantly with drain removal or no drainage, for at least 7 days, are allowed).
12. Participants with varices in the esophagus or stomach that require immediate intervention (e.g., ligation or sclerotherapy), or who are considered by the investigator or a gastroenterologist or hepatologist to be at high risk for bleeding, have evidence of portal hypertension (including splenomegaly on imaging), or have a history of variceal bleeding, must have endoscopic assessment within 3 months prior to the first start of study treatment.
13. Unhealed gastrointestinal obstruction, perforation, or fistula, or participants at risk of gastrointestinal obstruction or perforation (including but not limited to acute diverticulitis and abdominal abscess), or a history of extensive bowel resection (partial colectomy or extensive small bowel resection accompanied with chronic diarrhea), Crohn's disease, ulcerative colitis, or chronic diarrhea. Note: The digestive tract refers to the muscular tube from the oral cavity to the anal canal, including the oral cavity, pharynx, esophagus, stomach, small intestine (duodenum, jejunum, and ileum), large intestine (cecum, appendix, colon, and rectum), and anal canal.
14. After endoluminal stenting of the trachea and after stenting of the digestive tract, and the participant did not resume normal diet or defecation.
15. Participants with biliary obstruction, unless local treatment for obstruction (e.g., endoscopic stent placement or percutaneous liver drainage) has been performed and TBIL has decreased to less than 1.5 × ULN.
16. Hepatic encephalopathy, hepatorenal syndrome, or cirrhosis with Child-Pugh Class B or above.
17. Significant malnutrition, such as malnutrition requiring parenteral nutrition; except for those who have not used intravenous nutrition within 4 weeks before the first study treatment.
18. Uncontrolled active infection, including the following:

    1. Infection requiring systemic antibiotic, antiviral, or antifungal therapy.
    2. Human immunodeficiency virus (HIV) infection, or positive for HIV 1/2 Ab.
    3. Acute or chronic active hepatitis B, defined as hepatitis B surface antigen positive (regardless of the results of antibodies to other antigens) or hepatitis B core antibody positive only (hepatitis B surface antibody negative and hepatitis B e antibody negative), and hepatitis B virus (HBV) DNA ≥ 1 × 10 4 copies/mL or ≥ 2000 IU/mL; or acute or chronic active hepatitis C, defined as hepatitis C virus (HCV) antibody positive and HCV RNA titer above the lower limit of detection.
    4. Active tuberculosis infection, or still receiving anti-tuberculosis treatment, or received anti-tuberculosis treatment within 1 year before the first dose of study drug.
    5. Active syphilis infection or latent syphilis requiring treatment.
19. History of immunodeficiency diseases, including congenital or acquired immunodeficiency diseases.
20. History of allogeneic organ transplantation, allogeneic bone marrow transplantation, or autologous hematopoietic stem cell transplantation (except corneal transplantation).
21. Pregnant or lactating (may be considered if breastfeeding is discontinued) female participants, or participants planning to become pregnant.
22. Ineligible for any drug under study. Participants with contraindications to trastuzumab, pertuzumab monoclonal antibody, taxanes according to local prescribing information or IBI354 per the IBI354 Investigator's Brochure cannot be enrolled in the study.
23. Participant has known allergic or hypersensitivity reactions to the study treatments, camptothecin and its derivatives, other ADCs/anti-HER2 antibodies, and any excipients.
24. Complicated with other primary malignant tumors within 3 years or other malignant tumors with active or recurrent risk, excluding radically resected non-melanoma skin cancer (mainly including squamous cell carcinoma of skin and basal cell carcinoma of skin), radically resected carcinoma in situ, and papillary thyroid carcinoma.
25. Participation in any other interventional clinical study, except for observational (non-interventional) studies or follow-up period after the end of study treatment in interventional studies.
26. Presence of substance abuse (excessive or inappropriate use of drugs, alcohol, or other harmful substances that may lead to physical, psychological, or social problems) or other acute or chronic diseases or laboratory abnormalities that, in the opinion of the investigator, may interfere with the participant's participation in the clinical study, increase the risk of study participation or drug administration, interfere with the interpretation of study results, or render the participant unsuitable for participation in the study in the judgment of the investigator.
27. The participant has a neurologic, psychiatric, or psychological illness or social condition that would interfere with trial compliance, substantially increase the risk of adverse events, or prevent the participant from providing written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2026-02-28 (Estimated); Primary Completion 2028-04-28 (Estimated); Study Completion 2030-05-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) by Blinded Independent Central Review (BICR) assessment | Until progression or death, up to 54 months
  Defined as time from date of randomisation until the date of objective radiological disease progression according to Blinded Independent Central Review (BICR) using RECIST 1.1 or death by any cause.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) by Investigator assessment | Until progression or death, up to 54 months
  Defined as time from date of randomisation until the date of objective radiological disease progression according to Investigator using RECIST 1.1 or death by any cause.
Overall Survival (OS) | Until death, up to 54 months
  OS is defined as the time from randomisation until the date of death due to any cause.
Objective Response Rate (ORR) by BICR and Investigator assessment | Until progression or death, up to 54 months
  ORR is defined as the proportion of participants who have a complete response (CR) or partial response (PR) based on BICR and investigator assessment using RECIST 1.1.
Duration of Response (DoR) by BICR and Investigator Assessment | Until progression or death, up to 54 months
  DoR is defined as the time from date of first detection of objective response until the date of objective radiological disease progression according to BICR and investigator assessment using RECIST 1.1 or death in the absence of progression.
Disease control rate (DCR) by BICR and Investigator assessment | Until progression or death, up to 54 months
  DCR is defined as the proportion of participants in the analysis population achieving disease control (confirmed CR, PR, or stable disease [SD]) based on BICR and investigator assessment using RECIST 1.1.
Time to response (TTR) by BICR and Investigator assessment | Until progression or death, up to 54 months
  TTR is defined as the time from randomization to the first CR or PR among participants with confirmed ORR assessed by BICR and investigator per RECIST v1.1.
Safety and tolerability of IBI354, alone or with pertuzumab | Until progression or death, up to 54 months
  Number of AEs according to NCI-CTCAE Version 5.0 per each treatment arm
Immunogenicity of IBI354 | Until progression or death, up to 54 months
  Number and percentage of participants who develop anti-drug antibody (ADA) for IBI354

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China